CLINICAL TRIAL: NCT07168902
Title: A Phase 2 Evaluation of the Safety, Ocular Tolerability, and Efficacy of Topical Ophthalmic BL1107 Versus Timolol in Adults With Primary Open Angle Glaucoma or Ocular Hypertension
Brief Title: Phase 2 Study of BL1107 Eye Drops vs. Timolol in Adults With Primary Open Angle Glaucoma or Ocular Hypertension
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RX01-BL1107-1201
Record Dates: First submitted 2025-09-05; First posted 2025-09-11 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BL1107 Low dose (Experimental)
  Interventions: Drug: BL1107 Low dose
- BL1107 High dose (Experimental)
  Interventions: Drug: BL1107 High dose
- Timolol maleate 0.5% (Active Comparator)
  Interventions: Drug: Timolol maleate 0.5%

INTERVENTIONS:
Drug: BL1107 Low dose — Dosed twice daily for 28 days.
  Arms: BL1107 Low dose
Drug: BL1107 High dose — Dosed twice daily for 28 days.
  Arms: BL1107 High dose
Drug: Timolol maleate 0.5% — Dosed twice daily for 28 days.
  Arms: Timolol maleate 0.5%

SUMMARY:
Phase 2 Study of BL1107 Eye Drops vs. Timolol in Adults with Primary Open Angle Glaucoma or Ocular Hypertension

DETAILED DESCRIPTION:
This study will evaluate the safety and efficacy of BL1107 in adults with primary open-angle glaucoma or ocular hypertension in both eyes. This is a randomized, double-masked, parallel comparison to evaluate two concentrations of BL1107 in both eyes compared with timolol 0.5% for 28 days.

ELIGIBILITY:
Inclusion criteria:

* Ocular hypertension or primary open-angle glaucoma in each eye

Exclusion criteria:

* History of orthostatic hypotension
* Any active ocular disease
* Anticipated wearing of contact lenses during study
* Contraindication to pupil dilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2025-10-24 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in visual field mean deviation in the study eye at Day 28/Exit. | Assessed at Day 28

SECONDARY OUTCOMES:
Proportion of participants achieving ≥15-letter improvement in low-luminance best-corrected visual acuity (LL-BCVA) in the study eye at Day 28/Exit. | Assessed at Day 28
Proportion of participants achieving ≥10-letter improvement in low-luminance best-corrected visual acuity (LL-BCVA) in the study eye at Day 28/Exit. | Assessed at Day 28
Hour-matched change from Baseline in intraocular pressure (IOP) in the study eye at Day 28/Exit. | Assessed at Day 28

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Global Research Management, Inc., Glendale, California
  - Eye Research Foundation, Newport Beach, California
  - Levenson Eye Associates, Jacksonville, Florida
  - Central Florida Eye Associates, Lakeland, Florida
  - Lee Shettle Eye and Hearing, Largo, Florida
  - Andover Eye Associates, Andover, Massachusetts
  - Scott & Christie and Associates, PC, Cranberry Township, Pennsylvania
  - Total Eye Care, P.A., Memphis, Tennessee